CLINICAL TRIAL: NCT07155577
Title: Investigation of the Effects of Pes Planus Deformity on Gait Parameters at Different Inclines
Brief Title: Effects of Pes Planus on Gait at Different Inclines
Status: Recruiting | Type: Observational
Sponsor: Hacettepe University (Other)
Collaborators: Yuksek Ihtisas University (Other)
Responsible Party: Principal Investigator, Güngör Beyza ÖZVAR, Principal Investigator, Hacettepe University
Other Study IDs: Pes Planus
Record Dates: First submitted 2025-08-27; First posted 2025-09-04 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Flatfoot; Gait
MeSH Terms: conditions — Flatfoot

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Flexible Pes Planus Group: Adults aged 18-35 years with bilateral flexible pes planus, confirmed by Jack's toe-raise test and navicular drop ≥10 mm
- Healthy Control Group: Adults aged 18-35 years with normal BMI and no pes planus deformity.

SUMMARY:
This study aims to investigate the effects of pes planus deformity on gait spatiotemporal parameters and pelvic kinematics during walking on different inclines. Participants will include healthy adults aged 18-35 years with flexible bilateral pes planus and normal body mass index. Pes planus severity will be evaluated using the Jack's toe-raise test and the navicular drop test. Gait parameters such as walking speed, cadence, stride length, stance and swing phase percentages, gait cycle duration, as well as pelvic tilt, obliquity, and rotation symmetry will be measured using the BTS-G wireless sensor system. Assessments will be performed on both flat and inclined treadmill conditions. The findings are expected to provide new insights into the biomechanical adaptations of pes planus during walking and contribute to the development of an individualized rehabilitation protocol.

DETAILED DESCRIPTION:
This study will evaluate the effects of pes planus deformity on gait spatiotemporal parameters and pelvic kinematics during walking on flat and inclined surfaces. Flexible pes planus will be confirmed with Jack's toe-raise test, and severity will be assessed using the navicular drop test.

Healthy adults aged 18-35 years with bilateral flexible pes planus and normal BMI will be included. Exclusion criteria are lower extremity injury or surgery in the last 6 months, chronic ankle instability, other musculoskeletal disorders, or orthotic use.

Gait will be assessed with the BTS-G wireless sensor system, recording speed, cadence, stride length, stance and swing phase percentages, gait cycle duration, pelvic tilt, obliquity, and rotation symmetry. Participants will walk in standard sports shoes on level and inclined treadmill conditions. Data will be analyzed to determine biomechanical differences across surfaces.

The findings may provide insights into how pes planus influences gait and contributes to rehabilitation and footwear strategies.

ELIGIBILITY:
Inclusion Criteria: **Pes Planus Group

* Age 18-35 years
* Normal BMI
* Bilateral, asymptomatic flexible pes planus
* Navicular drop ≥10 mm (both feet)
* Willing and able to provide informed consent and complete the procedure.

  **Healthy Control Group
* Age 18-35 years
* Normal BMI
* No pes planus deformity; otherwise healthy and able to complete procedures

Exclusion Criteria:** both groups

* Use of orthotics/insoles
* Musculoskeletal disorders affecting gait (other than pes planus in the case group)
* Lower extremity injury or surgery within the last 6 months
* Chronic ankle instability
* Any treatment related to the lower extremity/pes planus within the last 6 months

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Adults aged 18-35 years with normal body mass index will be recruited. The study will include two groups:
  Flexible Pes Planus Group: Participants with bilateral, asymptomatic, flexible pes planus confirmed by Jack's toe-raise test and a navicular drop ≥10 mm.
  Healthy Control Group: Participants without pes planus deformity and with normal foot posture.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2026-01-25 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Gait Speed (Level vs. Inclined Walking) | up to 6 months
  Self-selected walking speed (m/s) measured during 20-m trials under level and inclined treadmill conditions using the BTS-G wireless sensor (L4-L5 placement). Between-group (pes planus vs control) and within-condition comparisons.
Cadence | up to 6 months
  Steps per minute captured by BTS-G during level and inclined walking; between-group and within-condition comparisons.Unit of Measure: steps/min.
Stride Length | up to 6 months
  Stride length (cm) during level and inclined walking recorded via BTS-G; between-group and within-condition comparisons.
Stance and Swing Phase Percentages | up to 6 months
  Percentage of the gait cycle spent in stance and swing (%) under level and inclined conditions using BTS-G; between-group and within-condition comparisons.
Pelvic Kinematics-pelvic tilt | up to 6 months
  Pelvic tilt recorded with BTS-G sensor across barefoot, 2 cm heel, and 6 cm heel conditions. It will be recorded as a degree.
Pelvic Kinematics-pelvic obliquity | up to 6 months
  Pelvic obliquity recorded with BTS-G sensor across barefoot, 2 cm heel, and 6 cm heel conditions. It will be recorded as a degree.
Pelvic Kinematics- pelvic rotation | up to 6 months
  Pelvic rotation recorded with BTS-G sensor across barefoot, 2 cm heel, and 6 cm heel conditions. It will be recorded as a degree.

SECONDARY OUTCOMES:
Navicular Drop (Severity of Pes Planus) | Baseline (prior to treadmill assessments)
  Navicular drop distance measured to quantify pes planus severity (baseline characterization).Unit of Measure: mm.
BMI (Body Mass Index) | Baseline (prior to treadmill assessments)
  Calculated as weight(kg)/height(m²) for baseline characterization.Unit of Measure: kg/m².

CONTACTS AND LOCATIONS:
Overall Officials: Aybuke Ertugrul, Principal Investigator — Yuksek Ihtisas University; Elıf Ceren Ersoy, Principal Investigator — Yuksek Ihtisas University; Busra Kalkan Balak, Study Director — Yuksek Ihtisas University; Zehranur Dağasar, Principal Investigator — Yuksek Ihtisas University
Locations (1):
- Yuksek Ihtisas University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No